CLINICAL TRIAL: NCT03362008
Title: A Randomized, Open-label, 2-Way, 2-Period, Single-Dose Crossover Clinical Study to Compare the Pharmacokinetic Characteristics and the Safety Between Zeropix Tablet 1 mg and Champix® Tablet 1 mg in Healthy Adult Male Subjects
Brief Title: Compare the Pharmacokinetic Characteristics and the Safety Between Zeropix and Champix in Healthy Adult Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JLP-1607-101-PK
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Smoking, Cigarette
MeSH Terms: conditions — Cigarette Smoking | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Period I: administration of Zeropix Period II: administration of Champix®
  Interventions: Drug: Zeropix; Drug: Champix®
- Group II (Experimental): Period I: administration of Champix® Period II: administration of Zeropix
  Interventions: Drug: Zeropix; Drug: Champix®

INTERVENTIONS:
Drug: Zeropix — administration of Zeropix
Drug: Champix® — administration of Champix®

SUMMARY:
This study is a randomized, open-label, 2-way, 2-period, single-dose crossover clinical study to compare the pharmacokinetic characteristics and the safety between zeropix tablet 1 mg and champix® tablet 1 mg in healthy adult male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male older than 19 to 45 years at the time of screening
2. Body weight more than 50kg and Body Mass Index(BMI) 18~29 kg/m2 ☞ BMI = (weight [kg])/(height [m])2 3. Subject judged to be eligible by physical examination and interview conducted according to the study protocol. Thus, Subject should not have congenital/chronic disease or pathological symptoms/findings

Exclusion Criteria:

1. Subject currently with or has a history of cardiovascular , respiratory, hepatic, renal, neurological, endocrine, hemato-oncology, psychiatric, urinary diseases that is clinically significant
2. Subject with a history of significant hypersensitivity or clinically significant hypersensitivity reaction to varenicline and other drugs (aspirin, antibiotic…etc.)
3. Systolic blood pressure ⩽100mmHg or ⩾ 150mmHg, diastolic blood pressure⩽55mmHg or ⩾ 95mmHg
4. Subject with a history of gastrointestinal disease (i.e. Crohn's disease, ulcer…etc.) or gastrointestinal surgery (not including, simple appendectomy or hernia surgery) that can affect drug absorption
5. Subject with the following results in the clinical laboratory tests

   * Aspartate Transaminase(AST) or Alanine Transaminase(ALT) > 2 x upper limit of normal range
   * Total Bilirubin > 2.0 mg/dl
   * CK > 2 x upper limit of normal range
   * eGFR < 60 mL/min/1.73m2
6. Subject who takes alcohol > 21 units/week, 1unit=10g=12.5ml of pure alcohol) or can't stop drinking during the clinical trials
7. Subject who smokes> 10 cigarettes/day or can't stop smoking during the clinical trials

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
AUCt of Varenicline | 96 hours
Cmax of Varenicline | 96 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No